CLINICAL TRIAL: NCT05493228
Title: the Role of Dexmedetomidine (Precedex) Infusion on Intraoperative Propofol & Fentanyl Requirements in Spine Surgery for Pediatric Cancer Patients
Brief Title: Dexmedetomidine Infusion on Intraoperative Propofol,Fentanyl Requirements in Spine Surgery for Pediatric Cancer Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Cancer Hospital Egypt 57357 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CCHE-BT005
Record Dates: First submitted 2022-08-01; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-06

CONDITIONS: Spine Cancer; Anesthesia
MeSH Terms: conditions — Spinal Cord Neoplasms | interventions — Dexmedetomidine; Sodium Chloride; Fluoridation

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, double-blinded clinical trial will be done on all included cases. They will be divided into two groups after induction of general anathesia using propofolwhich will be started at 100 ug/kg/min) and titrated to maintain the bispectral index at 40-60 and fentanyl will be started at 0.5ug/kg/min) and to be adjusted as needed to control the hemodynamic response to the surgical procedure and maintain the mean arterial pressure (MAP) at 55-65 mmHg. Then will randomly divided using Block Stratified Randomized Software program, after obtaining informed consent from eligible patient or his caregiver into two Arms:
  Arm A: will receive dexmedetomidine infusion at the rate of 0.5 μg kg-1 hr-1, started after the induction of general anesthesia without a loading dose which is colorless solution.
  Arm B :will receive placebo (saline injection) only after the induction of general anesthesia
Who Masked: Participant, Care Provider, Investigator
Masking Description: The PI (anesthesiologist), neurosurgeon ,patient, all assisting surgeons and anesthesiologist as well operating and circulating nurse will be blinded to the study arm to which patient belongs to. Only clinical trial unit and pharmacist will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient is receiving dexmedetomidine (Experimental): dexmedetomidine infusion at the rate of 0.5 μg kg-1 hr-1, started after the induction of general anesthesia without a loading dose
  Interventions: Drug: Precedex Injectable Product
- standard treatment (saline) (Placebo Comparator): saline injection only after the induction of general anesthesia
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Precedex Injectable Product — Precedex activates 2-adrenoceptors, and causes the decrease of sympathetic tone, with attenuation of the neuroendocrine and hemodynamic responses to anesthesia and surgery; it reduces anesthetic and opioid requirements; and causes sedation and analgesia. it is used before and/or during surgical
  Other Names: dexmedetomidine
  Arms: patient is receiving dexmedetomidine
Drug: Saline — mixture of sodium chloride (salt) and water in solution with 0.90% w/v of NaCl
  Other Names: Salt water
  Arms: standard treatment (saline)

SUMMARY:
The purpose of this trial is to investigate whether the effect of a low-dose dexmedetomidine infusion will decrease propofol consumption or not through a double blinded randomized controlled trial done in children cancer hospital 57357.

DETAILED DESCRIPTION:
Spinal surgery with instrumentation is associated with the risk of iatrogenic injuries to the spinal cord. The combination of somatosensory evoked potential (SSEP) and transcranial electric motor evoked potential (tcemep) monitoring has resulted in a high degree of sensitivity in predicting postoperative neurologic outcomes. Anesthetic agents have a dose-dependent adverse effect on the ability to record evoked potential responses. Many commonly used anesthetic agents produce a dose-dependent amplitude reduction and latency prolongation of evoked responses, which may impair diagnosis of intraoperative spinal cord injury. Neuroprotection is the cornerstone of anesthetic management in neurosurgery. Preserving the quality of SSEP and motor evoked potential (MEP) and minimizing the effects of anesthetic agents on neurologic monitoring are thus investigators' priorities.

Motor-evoked potential (MEP) and somatosensory-evoked potential (SSEP) monitoring are universally used during spine surgeries, which poses risks to the functional integrity of descending motor and ascending sensory pathways.

MEP baseline recording is obtained at the start of surgery determining the amplitude. The alarming criteria for MEP are attenuation of more than 50 % in motor response amplitude for segmental tcMEP, more than 80 % for long tract tcMEP and/or abolishment of tcMEP data. Any significant change is immediately reported to the surgeons.

Prior to skin incision, SSEP baseline amplitude and latency of cortical potential peaks were recorded (N20 for upper SSEP and P37 for lower SSEP). The alarming criteria of SSEP are 50% decreased amplitude and/or more than 10% increased latency compared to baseline.

The anesthetic agents have effects on the latency and amplitude of MEP and SSEP monitoring which is dose-dependent. Total intravenous anesthesia (TIVA) with propofol and opioid is commonly recommended for surgeries that require MEP and SSEP monitoring. However, propofol administered with a large dose affects MEP monitoring.

Using dexmedetomidine has the ability of sparing hypnotics usage, especially propofol, thus facilitating MEP and SSEP monitoring with providing its beneficial effects.

The addition of dexmedetomidine (0.5 μg/kg loading dose infused over 10 min followed by a constant infusion rate of 0.5 μg/kg/h) to propofol-remifentanil regimen does not exert an adverse effect on MEP and SSEP monitoring in adult patients undergoing thoracic spinal cord tumor resection and the addition of dexmedetomidine reduces the propofol requirements for a comparable BIS measurement. Another study that supports this regimen concluded that SEPs and MEPs were maintained in the patients who are administered with the dexmedetomidine etomidate fentanyl combined anesthesia during spinal surgery. Also, it was find that dexmedetomidine changes SSEP amplitude at clinically nonsignificant levels and may be safely used in intraoperative nerve monitoring at up to 1.2mg/ kg/h .

The most attractive form of display for the calculated power spectrum during anaesthesia is the compressed spectral array (CSA), where the component power is plotted as a function of frequency for each analysed epoch. Power spectrum analysis and subsequent display of data in the CSA format provide a simplified identification of small changes in a complex EEG.

Total intravenous anesthesia (TIVA) with propofol and opioid is commonly recommended for surgeries that require MEP and SSEP monitoring. However, even propofol used with a large dose can also affect MEP monitoring. Despite its efficacy, dose-related adverse effects may occur with propofol including prolonged awakening times, lipemia, and alteration of platelet function. Additionally, although more of a concern with its prolonged use in the ICU setting, recent attention has focused on the potential development of the 'propofol infusion syndrome' during intraoperative care.

Dexmedetomidine, an alpha 2-receptor agonist, is routinely used to provide analgesia and sedation without respiratory depression in critically ill patients. Its hemodynamic stability, negligible respiratory depression, and reduction of other anesthetic and analgesic requirements make it an interesting option for intraoperative use as an adjunctive agent for general anesthesia .When dexmedetomidine is added to a propofol infusion, it decreases the dose of propofol required,provides moderate hypotension, decreases blood loss, and allows monitoring of MEPs and SSEPs. The dose of dexmedetomidine often quoted in the literature is a bolus of 1 μg kg-1 hr-1 over 10 min followed by infusion of 0.2-0.7 μg kg-1 hr-1, but this dose frequently results in bradycardia and hypotension. Recently,this study is planned to evaluate the effects of intraoperative IV infusion of a low-dose (0.5 μg kg-1 hr-1) dexmedetomidine in patients undergoing spine surgery.

Researchers have administered an intraoperative continuous infusion of lower doses of dexmedetomidine without a prior bolus.

ELIGIBILITY:
Inclusion Criteria:

* spinal cord tumor resection based on magnetic resonance imaging (MRI) studies.
* age between 5 -18 years old
* American Society of Anesthesiologists (ASA) physical status II or III.

Exclusion Criteria:

* Emergency spine surgery
* Cardiac patients
* Any individual with stage 4 or greater chronic kidney disease (eGFR< 30 ml/min) and/or requiring dialysis
* liver failure defined as a history of cirrhosis or fulminant hepatic failure
* Preoperative dexmethatodine use
* Preoperative systolic hypertension defined by a systolic blood pressure greater than 130 mmHg in the surgical admission suite
* Enrolled in another study within 30 days.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2023-04-17 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Rate of propofol infusion per hour | during surgery
  measured by infusion pump in ml/hr
Change in MEP amplitude and latency | at baseline and during surgery
  intraoperatively monitoring by neurophysiology in MV
Depth of anesthesia by bispectral index | during surgery
  intraoperatively by anesthesiologist BIS within normal range 40-60
change in SSEP amplitude and latency | at baseline and during surgery
  intraoperatively monitoring by neurophysiology in MV

SECONDARY OUTCOMES:
to access rapid recovery in both arms | immediately after surgery
  To access whether using dexmedetomidine infusion will affect time of recovery
to access the event of hypotension in both arms | baseline ,during surgery and immediately after surgery
  will measured by blood pressure (mmHg)
to access the event of bradycardia in both arms | baseline, during surgery and immediately after surgery
  will measured by Heart rate (beat/min)

CONTACTS AND LOCATIONS:
Overall Officials: suzan m Adlan, MD, Principal Investigator — 57357 children cancer hospital
Locations (1):
- Children's Cancer Hospital Egypt 57357 Cairo, Egypt, Cairo, Egypt